CLINICAL TRIAL: NCT04723992
Title: 25-Year Experience With Polytraumatized Patients in a Level 1 Trauma Center.: Polytrauma Between 1995 and 2019: What Has Changed
Brief Title: 25-Year Experience With Polytraumatized Patients in a Level 1 Trauma Center
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Valerie Weihs, Principle Investigator, Medical University of Vienna
Other Study IDs: 1146/2020
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective analysis — The investigators retrospectively analyzed the outcome and possible prognostic factors in polytrauma patients.

SUMMARY:
In this study patients who were admitted to our hospital with critical injuries were enrolled retrospectively from January 1992 to December 2019. Patients with an ISS>16 points, an AIS >3 in one body region and at least 2 different body regions affected were included. Possible prognostic factors were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ISS >16 points
* AIS >3 in one body region
* at least 2 body regions affected

Exclusion Criteria:

* patients younger than 18 years of age
* isolated traumatic brain injury
* minor injuries (AIS <3 or ISS <16 points)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of polytrauma patients.
Sampling Method: Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 1992-01; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality in polytrauma patients. | January 1st 1992 to December 31st 2019
Possible prognostic factors influencing the outcome of polytrauma patients. | January 1st 1992 to December 31st 2019
  Evaluation of concomitant traumatic brain injury, resuscitation, injury severity and trauma mechanisms in polytrauma patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Traumatology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weihs V, Frenzel S, Dedeyan M, Hruska F, Staats K, Hajdu S, Negrin LL, Aldrian S. 25-Year experience with adult polytraumatized patients in a European level 1 trauma center: polytrauma between 1995 and 2019. What has changed? A retrospective cohort study. Arch Orthop Trauma Surg. 2023 May;143(5):2409-2415. doi: 10.1007/s00402-022-04433-1. Epub 2022 Apr 12. PMID 35412071